CLINICAL TRIAL: NCT02233608
Title: A Randomized Pilot Study of Conventional Versus Advanced Pelvic Floor Exercises to Treat Urinary Incontinence After Radical Prostatectomy
Brief Title: Advanced Pelvic Floor Training Program for Prostate Cancer Surgery
Acronym: AFPX
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Guelph-Humber (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Daniel Santa Mina, Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D2014-20
Record Dates: First submitted 2014-09-03; First posted 2014-09-08 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy
Keywords: Prostate cancer; Radical prostatectomy; Pelvic floor muscle exercises; Pfilates; Hypopressives; Urinary Incontinence
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): The usual care group will receive generic pelvic floor muscle exercise (PMFX) instructions and demonstrations by the research coordinator at the initial post-operative time point. This will include instruction on how to engage the pelvic floor and specific PFMX prescription. Repetition volume will start at 20 repetitions per day during weeks 1-2; 60/day during weeks 3-4; and 90/day during weeks 5-6, and 100+/day for weeks 7-26. The total number of repetitions will be divided equally between rhythmic (contract and relaxed over one second) and sustained contractions (contract and hold for up to 10 seconds).
- Advanced Pelvic Floor Exercise (APFX) (Experimental): Participants in this group will receive detailed week-by-week description of the program. The program progresses participants through stages of training every two weeks, starting the introduction of basic PFMX, and slowly incorporates Pfilates and Hypopressives exercises until week 8, where patients will maintain the final stage of training until week 26 or urinary incontinence is completely resolved.
  Interventions: Behavioral: Advanced Pelvic Floor Muscle Exercise (APFX)

INTERVENTIONS:
Behavioral: Advanced Pelvic Floor Muscle Exercise (APFX)
  Arms: Advanced Pelvic Floor Exercise (APFX)

SUMMARY:
Radical prostatectomy is a common and effective treatment for prostate cancer but is associated with urinary incontinence that can persist for several months after surgery and significantly reduce quality of life. Studies have shown that routine performance of pelvic floor exercises after radical prostatectomy can aid in the recovery of urinary control; however, conventional pelvic floor exercises do not produce consistent results. Research indicates that incorporating other deep abdominal muscles can further activate the pelvic floor making it stronger than by activating the pelvic floor alone. Specifically, 'Pfilates' and 'Hypopressives' are two new techniques that combine traditional pelvic floor exercises with activation of supportive muscles. Our proposed study will be the first to test the effect of an advanced pelvic floor exercise training program that includes Pfilates and Hypopressives to treat urinary incontinence following radical prostatectomy. Our primary aim of this study is to assess the feasibility of conducting a full-scale RCT of an advanced pelvic floor exercise training program, including standard pelvic floor exercises, Pfilates, and Hypopressives techniques on urinary incontinence. Feasibility will be determined by measuring recruitment success, retention, outcome capture, and intervention adherence, tolerance, and safety. We hypothesize men under going radical prostatectomy for prostate cancer in the advance pelvic floor training program will report greater improvement in urinary incontinence and health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men with localized prostate cancer (stage cT1-cT2) who have consented for radical prostatectomy (open retropubic, laparoscopic, robot-assisted laparoscopic)
* Between the the ages of 40 and 80 years
* Proficient in English

Exclusion Criteria:

* i) Diagnosed with a known neurological disease, autoimmune connective tissue disorder;
* ii) Have prior experience with pelvic floor training by a healthcare provider;
* iii) Have uncontrolled hypertension;
* iv) Have diagnosed COPD (Chronic Obstructive Pulmonary Disease) and/or chronic restrictive respiratory disease; or
* v) Have a history of inguinal herniation

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-09-28 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Recruitment | When recruitment is complete (approximately 12 months after study initiation; October 2015)
  Prior pelvic floor training trials in prostate cancer patients undergoing radical prostatectomy have observed recruitment rates of 21-70%. We will measure recruitment success through participant recruitment per week and record reasons for non-participation from those who inquire about the study and are eligible to participate but refuse.
Adherence to intervention group | 26 weeks post-operatively
  Adherence to the two groups (standard pelvic floor exercises and advanced pelvic floor exercises) will be measured through a logbook that is included in their respective program manuals as well as a logbook completed by the research coordinator during the weekly telephone communications.
Study retention | 26 weeks post-operative
  Retention will be assessed by measuring attrition throughout the intervention period and at each assessment.
24-hour Pad Test for Urinary Leakage | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 weeks post-operatively
  A 24-hour pad test will be used to measure urinary incontinence by assessing the quantity of urine lost in one day. A urinary leakage pad is measured after a 24-hour period and compared to the unused pad weight and is used to most accurately assess the severity of urinary incontinence.
Pelvic Floor Strength | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26, weeks post-operatively
  Digital rectal examination of pelvic floor strength by a specially trained pelvic floor physiotherapist will be conducted. Pelvic floor strength will be graded on the Modified Oxford Scale.

SECONDARY OUTCOMES:
Quality of Life | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 weeks post-operative
  Prostate specific quality of life will be measured using the Functional Assessment of Cancer Treatment-Prostate (FACT-P) and the Patient-Oriented Prostate Utility Scale (PORPUS).
3-Day Bladder Diary for Urinary Incontinence | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 week post-operatively
  The bladder diary is a standard instrument for self-reporting voiding patterns. Items include fluid intake, frequency of toilet voids, episode of urine loss, number of pads used, and activity during event for the three-day period. Bladder diaries are widely used in clinical trials assessing urinary incontinence after radical prostatectomy.
Self-Reported Urinary Incontinence, Prostate Symptoms, and Erectile Function | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 week post-operatively
  Urological symptoms are assessed using the International Prostate Symptom Score (IPSS). Additional, a single item regarding leaking urine and bladder control from the PORPUS will be used to evaluate incontinence. Erectile function will be assessed using the 5-item International Index of Erectile Function scale (5-IIEF).
Body Composition | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 week post-operatively
  Body composition will be assessed via bioelectrical impedance analysis, height, weight, waist and hip circumference, and body mass index.
Physical Activity | At baseline, approximately 1 week prior to surgery, and 2, 6, 12, 26 weeks post-operatively
  Physical activity level will be measured wight he 3-item Godin Leisure Time Exercise Questionnaire - Leisure Score Index (GLTEQ-LSI).

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Santa Mina D, Au D, Alibhai SM, Jamnicky L, Faghani N, Hilton WJ, Stefanyk LE, Ritvo P, Jones J, Elterman D, Fleshner NE, Finelli A, Singal RK, Trachtenberg J, Matthew AG. A pilot randomized trial of conventional versus advanced pelvic floor exercises to treat urinary incontinence after radical prostatectomy: a study protocol. BMC Urol. 2015 Sep 16;15:94. doi: 10.1186/s12894-015-0088-4. PMID 26377550